CLINICAL TRIAL: NCT02696941
Title: SGLT2 Inhibitors and Metformin on Metabolism and Non-Alcoholic SteatoHepatitis
Acronym: SMASH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11693
Record Dates: First submitted 2016-02-12; First posted 2016-03-02 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Metformin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Participants with insulin resistance who have not yet started any diabetic medication will be recruited and will be prescribed metformin at standard clinical doses.
  Interventions: Drug: Metformin
- SGLT2 (Experimental): Participants with poorly controlled type 2 Diabetes (T2DM) who have been recommended to start an SGLT2 inhibitor will be recruited.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: Metformin — Metformin 500mg once daily and titrated weekly to a dose of 1000mg twice daily for 3 months
  Arms: Metformin
Drug: SGLT2 inhibitor — SGLT2 inhibitor has been recommended to be started as part of routine clinical care
  Arms: SGLT2

SUMMARY:
SGLT2 inhibitors have been proven to be effective in several preclinical rodent models of non-alcoholic fatty liver disease (NAFLD). Using a choline deficient diet to recapitulate some of the histological features of human non-alcoholic steatohepatitis (NASH), it was found that 5 weeks of SGLT2 inhibition led to significant reductions in hepatic triglyceride content and improved markers of liver fibrosis. Similarly, 4 weeks of treatment in obese mice led to improved glucose tolerance, reduced hepatic steatosis and reduced markers of liver oxidative stress in a dose dependent manner. These findings corresponded with an improvement in traditional liver function tests including the aminotransferases (ALT and AST). The widely used antidiabetic agent metformin has been shown in rodent models to increase hepatic insulin sensitivity and lower liver fat content which is in contrast to the findings in humans where metformin increases hepatic insulin sensitivity, reduces body weight but does not decrease liver fat content. The reason for the discrepancy between the animal and human studies, with regards to liver fat content remains unclear.

The investigators hypothesise the following:

* SGLT2 Inhibitors have the potential to decrease lipid accumulation in the liver through reduced de novo lipogenesis (DNL)
* There will be no decrease in endogenous lipid synthesis (DNL) with metformin and thus no change in liver fat content.

There are two arms to this study.

* Arm 1: x10 participants with poorly controlled type 2 Diabetes (T2DM) who have been recommended to start an SGLT2 inhibitor called dapagliflozin will be recruited.
* Arm 2: x13 participants with insulin resistance who have not yet started any diabetic medication will be recruited and will be prescribed metformin at standard clinical doses.

The two arms will run in parallel and all participants will undergo identical investigations before and after 3 months of treatment with either dapagliflozin or metformin. Investigations will include liver magnetic resonance imaging/spectroscopy, fat biopsy, fat microdialysis sampling, two-step hyperinsulinaemic euglycaemic clamp, breath sampling and stable glucose and palmitate isotope infusions.

The investigators aim to show that SGLT2 inhibition decreases liver fat whereas we aim to demonstrate why liver fat remains unchanged in humans, treated with metformin. These data will provide the first evidence for the use SGLT2 inhibitors in NAFLD, and will be highly informative for the design of future clinical studies. Moreover, the data gained from the metformin arm of the study will provide the first mechanistic evidence in humans of the effects of metformin on hepatic fatty acid metabolism.

ELIGIBILITY:
Inclusion Criteria:

Arm 1: SGLT2 inhibitors

* Volunteers with diagnosis of Type 2 Diabetes on oral anti-diabetic therapy at a stable dose for ≥3 months including one of the following:

  i. Metformin monotherapy ii. Sulphonylurea monotherapy iii. Metformin and Sulphonylurea dual therapy
* All volunteers will be due to start SGLT2 inhibitor therapy for inadequate glycaemic control and it will be prescribed according to licensed indications.

Arm 2: metformin

• Insulin resistant treatment naive individuals as defined by fasting insulin and / or glucose in top 10th percentile

Both arms:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 years and 70 years.
* BMI: 25-45 kg/m2
* HbA1C: 42-86mmol/mol
* Normal renal function

Exclusion Criteria:

Arm 1: SGLT2 inhibitors Volunteers taking insulin, glucagon-like peptide 1 analogues, thiazolidinediones, or dipeptidyl peptidase IV inhibitors

Arm 2: metformin Volunteers taking insulin, glucagon-like peptide 1 analogues, thiazolidinediones, SGLT2 inhibitors, metformin or dipeptidyl peptidase IV inhibitors

Both arms

* Age <18 or >70 years
* Body mass index <25 or >45kg/m2
* A blood haemoglobin <120mg/dL
* History of alcoholism or a greater than recommended alcohol intake (Recommendations > 21 drinks on average per week in men and > 14 drinks on average per week in women)
* Pregnant or nursing mothers
* History of severe claustrophobia
* Presence of metallic implants, pacemaker
* Haemorrhagic disorders
* Anticoagulant treatment
* History of albumin allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis | 3 months
  Liver fat measured by magnetic resonance imaging / spectroscopy (MRI/S)

SECONDARY OUTCOMES:
% contribution of newly synthesised lipid to circulating triglyceride levels | 3 months
  deuterated water incorporation into palmitate
Global insulin sensitivity | 3 months
  two-step hyperinsulinaemic-euglycaemic clamp
Hepatic insulin sensitivity | 3 months
  two-step hyperinsulinaemic-euglycaemic clamp
Intrabdominal fat | 3 months
  Intrabdominal fat depot measured at level of L4-L5, visible on liver MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy W Tomlinson, MD PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Marjot T, Green CJ, Charlton CA, Cornfield T, Hazlehurst J, Moolla A, White S, Francis J, Neubauer S, Cobbold JF, Hodson L, Tomlinson JW. Sodium-glucose cotransporter 2 inhibition does not reduce hepatic steatosis in overweight, insulin-resistant patients without type 2 diabetes. JGH Open. 2019 Nov 5;4(3):433-440. doi: 10.1002/jgh3.12274. eCollection 2020 Jun. PMID 32514450